CLINICAL TRIAL: NCT07265336
Title: Comparison of Base Excess in Arterial Blood Gases Between Patients With Severe Preeclampsia and Normotensive Pregnant Patients
Brief Title: Excess Base Comparison Between Pregnant Subjects With Severe Preeclampsia vs. Normotensive Pregnant Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head of Research Department, Saint Thomas Hospital, Panama
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4558
Record Dates: First submitted 2025-08-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Preeclampsia; Severe Preeclampsia
Keywords: Excess base; Severe preeclampsia; Arterial blood gases
MeSH Terms: conditions — Pre-Eclampsia | interventions — Blood Gas Analysis

STUDY DESIGN:
Intervention Model Description: Both groups will have a blood sample taken for arterial blood gases. This test is not always indicated in severe preeclampsia and very rarely in normal patients. This is he reason we consider the study interventional.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe preeclampsia (Experimental): Pregnant subjects with severe preeclampsia
  Interventions: Diagnostic Test: Arterial Blood gases
- Normotensive (Experimental): Pregnant subjects with normal blood pressure
  Interventions: Diagnostic Test: Arterial Blood gases

INTERVENTIONS:
Diagnostic Test: Arterial Blood gases — Determination of Excess Base in arterial blood gases before delivery / termination of pregnancy

SUMMARY:
The study's primary goal is to compare the base excess (BE) values-an indicator of metabolic changes-in two groups of patients at Santo Tomás Hospital: those with severe preeclampsia and healthy, pregnant individuals. Researchers will measure these values using an arterial blood gas test before delivery or surgery.

This is a prospective cohort study. The researchers will analyze various blood gas parameters, including pH, lactate, and BE, and then correlate the BE values with clinical variables and negative maternal outcomes.

The expected outcome is that a abnormal BE values will be linked to a greater severity of preeclampsia. If this association is confirmed, BE could serve as an additional marker for predicting the severity of the condition and may lay the groundwork for future research on diagnostic and therapeutic standards based on blood gas analysis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age: 24-40 weeks
* Cases: Diagnosis of severe preeclampsia
* Control: Normal blood pressure

Exclusion Criteria:

* Metabolic conditions that could hinder the results (diabetic ketoacidosis, sepsis, renal failure).
* Clinical conditions that could hinder the results (diarrhea, vomit)
* Recent use of bicarbonate

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Value of excess base | Immediately before delivery
  Total measure of excess base measured by gasometry in an arterial blood sample
Hypertensive crisis | From admission to day three (3) after delivery
  Elevation of the blood pressure above 160 (systolic) and 110 (diastolic).

SECONDARY OUTCOMES:
Lactate | Immediately before delivery
  Concentration of lactate measured by gasometry in a sample of arterial blood.
Bicarbonate | Immediately before delivery
  Concentration of bicarbonate measured by gasometry in arterial blood gases

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Study Chair — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Hospital, Panama City, Provincia de Panamá, Panama

IPD SHARING:
Plan to Share IPD: No